CLINICAL TRIAL: NCT02462603
Title: A Phase 2A Safety and Biomarker Study of EPI-589 in Mitochondrial Subtype and Idiopathic Parkinson's Disease Subjects
Brief Title: Safety and Biomarker Study of PTC-589 in Participants With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edison Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI589-15-002
Record Dates: First submitted 2015-05-20; First posted 2015-06-04 (Estimated); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; PD; EPI-589; EPI589
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTC589 (Experimental): Participants with Parkinson's disease (idiopathic and mitochondrial genetic subtype participants) will receive PTC589 at a dose of 500 milligrams (mg) (2 tablets of 250 mg each) orally twice daily (BID) for up to 3 months unless discontinued for safety or tolerability issues.
  Interventions: Drug: PTC-589

INTERVENTIONS:
Drug: PTC-589 — PTC-589 is a redox active molecule and will be provided in a 250 mg tablet formulation.
  Other Names: (R)-Troloxamide quinone

SUMMARY:
Open-label study with 30-day run-in phase and adaptive design component to include more participants if deemed appropriate by investigators.

DETAILED DESCRIPTION:
This is a within-subject, controlled open-label study seeking to determine if PTC-589 can alter the biochemical signature of Parkinson's disease as assessed by peripheral blood biomarkers, central nervous system (CNS) biomarkers, and urine biomarker analysis. In addition, data on a number of disease-relevant clinical measures will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr stage ≤3.0
* Ambulatory with or without assistance
* Sexually active fertile participants and their partners must agree to use medically accepted methods of contraception (such as, hormonal methods, including oral, subcutaneous, and intrauterine; barrier methods, including male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 3 months after the last dose of study treatment.
* Willingness and ability to comply with study procedures
* If on medications for Parkinson's disease drugs, then medication regimen must be stable for 60 days prior to enrollment
* Abstention from use of other investigative or non-approved drugs for the duration of the trial

For Idiopathic Participants

* A diagnosis of idiopathic Parkinson's disease confirmed by the presence of bradykinesia plus one or both of the following symptoms: rigidity or resting tremor; and with an abnormal DaTscan consistent with a dopaminergic deficit
* Age 40 to 75 years
* Within 5 years of diagnosis of Parkinson's disease

For Genetic Subtype Participants

* A confirmed diagnosis of Parkinson's disease plus a genetic diagnosis consistent with Parkinson's disease, specifically PTEN-induced kinase 1 (PINK1), parkin, Leucine-rich repeat kinase 2 (LRRK2) or other mitochondrial genetic subtype
* Age 21 to 75 years

Exclusion Criteria:

* Allergy to PTC-589 or other components of the PTC-589 tablet formulation
* Use of antioxidant supplements, specifically vitamins E and C beyond the recommended daily allowance
* Other Parkinsonian disorders
* Montreal Cognitive Assessment (MoCA) score of <24
* Revised Hamilton Rating Scale for Depression ≥11
* Parkinsonism due to drugs or toxins
* Diagnosis of any other clinically significant neurologic disease that will confound the assessment of effect of study drug on disease progression
* Malignancy within past 2 years
* Pregnant or plans to become pregnant or breast feeding
* History of stroke
* History of brain surgery
* Hepatic insufficiency with liver function tests (LFTs) >3 times upper limit of normal
* Renal insufficiency as defined by creatinine >1.5 times normal
* End stage cardiac failure
* Participation within past 3 months and for duration of study in a trial of a device, drug, or other therapy for Parkinson's disease

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Klein, MD FACS, Study Director — Edison Pharmaceuticals
Locations (5):
- United States (3):
  - Cedar's Sinai, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
- DZNE Site, Tübingen, Germany
- University College of London,Dept. of Clinical Neuroscience, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- PTC589: Participants with Parkinson's disease (idiopathic and mitochondrial genetic subtype participants) received PTC589 at a dose of 500 milligrams (mg) (2 tablets of 250 mg each) orally twice daily (BID) for up to 3 months unless discontinued for safety or tolerability issues.
Period: Overall Study
Arm/Group | PTC589
Started | 44
Received at Least 1 Dose of Study Drug | 41
EITT Population (participant who received at least 1 dose of PTC589 and had a minimum of Month 3 assessment.) | 40
Completed | 40
Not Completed | 4
Not completed — Investigator Decision | 1
Not completed — Non-Compliance | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Safety population included any participant who received at least 1 dose of PTC589.
Groups:
- PTC589: Participants with Parkinson's disease (idiopathic and mitochondrial genetic subtype participants) received PTC589 at a dose of 500 mg (2 tablets of 250 mg each) orally BID for up to 3 months unless discontinued for safety or tolerability issues.
Arm/Group | PTC589
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-Related Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 4 months)
Population: Safety population included any participant who received at least 1 dose of PTC589.
Measure: Count of Participants; unit: Participants
Arm/Group | PTC589
Number analyzed (Participants) | 41
Participants | 0

2. Secondary Outcome: Change From Baseline in Movement Disorder Society Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Score at Month 3
Description: The MDS-UPDRS is a tool for monitoring the impact of Parkinson's disease, the degree of disability caused, and complications from treatment. Part I (13 items) evaluates nonmotor experiences of daily living (nM-EDL); Part II (13 items) evaluates motor experiences of daily living (M-EDL; Part III (18 items) is a motor examination; Part IV (6 items) examines motor complications (for example, motor fluctuations and dyskinesias). Each item was rated on a 5-point scale, ranging from 0 (normal) to 4 (severe), with higher score indicating greater severity and more impairment. Total score for Part I (nM-EDL) and Part II (M-EDL) each ranges from 0-52; for Part III (motor examination) ranges from 0-72; and for Part IV (motor complications) ranges from 0-24; with higher scores in each range for all 4 parts reflecting greater severity.
Time Frame: Baseline, Month 3
Population: Efficacy intent-to-treat (EITT) population included any participant who received at least 1 dose of PTC589 and had a minimum of the Month 3 assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTC589
Number analyzed (Participants) | 40
units on a scale
  nM-EDL Total Score: Baseline | 5.0 (4.51)
  nM-EDL Total Score: Change at Month 3 | -0.1 (3.93)
  M-EDL Total Score: Baseline | 5.8 (4.13)
  M-EDL Total Score: Change at Month 3 | 0.1 (3.54)
  Motor Examination Total Score: Baseline | 22.5 (8.60)
  Motor Examination Total Score: Change at Month 3 | -0.6 (6.72)
  Motor Complications Total Score: Baseline | 1.3 (2.34)
  Motor Complications Total Score: Change at Month 3 | -0.1 (2.17)

3. Secondary Outcome: Change From Baseline in Non-motor Symptoms Scale (NMSS) Total Score at Month 3
Description: Non-motor symptoms were evaluated using the NMSS which was divided into 30 questions in 9 different domains including such symptoms as dribbling saliva, constipation, depression, sleep disorders, apathy, hallucinations and dementia. Symptoms were quantified based on their severity (using a scale of 0 [none] to 3 [severe]) and frequency (using a scale of 0 [rarely] to 4 [very frequent]). Total score derived from adding up the product of the frequency score times severity score for each of the 30 questions. Total score ranged from 0 to 360, with a lower score indicating fewer symptoms.
Time Frame: Baseline, Month 3
Population: EITT population included any participant who received at least 1 dose of PTC589 and had a minimum of the Month 3 assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTC589
Number analyzed (Participants) | 40
units on a scale
  Baseline | 15.7 (14.84)
  Change at Month 3 | -0.6 (14.79)

4. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire - 39 (PDQ-39) Score at Month 3
Description: The PDQ-39 is a self-administered questionnaire for participants with Parkinson's disease that has 39 questions grouped in 8 dimensions: mobility (items 1-10), activities of daily living (items 11-16), emotional well-being (items 17-22), stigma (items 23-26), social support (items 27-29), cognitions (items 30-33), communication (items 34-36), and bodily discomfort (items 37-39). Each item was scored on a 5-point Likert scale (0 to 4) to indicate the frequency of each event; 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, and 4 = always or cannot do at all. Each dimension's total score ranged from 0-100, with lower scores indicating better health, and higher scores indicating more severe symptoms.
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTC589
Number analyzed (Participants) | 40
units on a scale
  Mobility: Baseline | 7.06 (12.543)
  Mobility: Change at Month 3 | 0.19 (7.281)
  Activities of daily living: Baseline | 11.56 (10.096)
  Activities of daily living: Change at Month 3 | 0.21 (10.676)
  Emotional well-being: Baseline | 10.84 (11.387)
  Emotional well-being: Change at Month 3 | 0.10 (10.180)
  Stigma: Baseline | 15.96 (17.685)
  Stigma: Change at Month 3 | -0.94 (16.602)
  Social support: Baseline | 1.88 (4.811)
  Social support: Change at Month 3 | 3.12 (9.750)
  Cognition: Baseline | 9.70 (12.085)
  Cognition: Change at Month 3 | -1.24 (8.747)
  Communication: Baseline | 6.25 (9.388)
  Communication: Change at Month 3 | 1.25 (10.777)
  Bodily discomfort: Baseline | 16.87 (15.390)
  Bodily discomfort: Change at Month 3 | 0.01 (14.501)

5. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension (EQ-5D) Score at Month 3
Description: EQ-5D is a questionnaire designed to provide measures of health-related quality of life states, consisting of 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has a 3 point response scale designed to indicate the level of the problem: 1 = no problems, 2 = some problems, 3 = extreme problems. A higher score indicated an increase in the level of problem. The EQ-5D also contains a visual analog scale (EQ-VAS), which records the respondent's self-rated health status on a vertical graduated visual analog scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). Higher score indicated improvement.
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTC589
Number analyzed (Participants) | 40
units on a scale
  Mobility: Baseline | 1.2 (0.36)
  Mobility: Change at Month 3 | 0 (0.36)
  Personal Care: Baseline | 1.1 (0.27)
  Personal Care: Change at Month 3 | 0 (0.36)
  Usual Activities: Baseline | 1.2 (0.42)
  Usual Activities: Change at Month 3 | 0.1 (0.35)
  Pain/Discomfort: Baseline | 1.3 (0.47)
  Pain/Discomfort: Change at Month 3 | 0.2 (0.48)
  Anxiety/Depression: Baseline | 1.1 (0.27)
  Anxiety/Depression: Change at Month 3 | 0.2 (0.50)
  VAS Score: Baseline | 81.0 (12.00)
  VAS Score: Change at Month 3: number analyzed (Participants) | 39
  VAS Score: Change at Month 3 | -1.9 (8.68)

6. Secondary Outcome: Montreal Cognitive Assessment (MoCA) Score
Description: MoCA is a 30-point questionnaire for cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Scores on the MoCA range from 0-30 with 26-30 indicating normal global cognition; 18-25 mild cognitive impairment; 10-17 moderate cognitive impairment; and <10 severe cognitive impairment.
Time Frame: Month 3
Population: EITT population included any participant who received at least 1 dose of PTC589 and had a minimum of the Month 3 assessment. Here, 'Number analyzed' signifies participants with normal, mild, moderate, or severe cognition impairment. Data for a specific severity level was not collected if no evaluable participants were available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTC589
Number analyzed (Participants) | 40
units on a scale
  Normal global cognition: number analyzed (Participants) | 33
  Normal global cognition | 28.5 (1.25)
  Mild cognitive impairment: number analyzed (Participants) | 7
  Mild cognitive impairment | 23.4 (1.40)
  Moderate cognitive impairment: number analyzed (Participants) | 0
  Severe cognitive impairment: number analyzed (Participants) | 0

7. Secondary Outcome: Beck Depression Inventory (BDI) Score
Description: The BDI is a self-reporting 21-item scoring tool that measures characteristic attitudes and symptoms of depression, including physical symptoms. Each of the 21 items on BDI tool represent a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 (symptom is absent) to 3 (symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items, which are interpreted as follows 1-10 (normal); 11-16 (mild mood disturbance); 17-20 (borderline clinical depression); 21-30 (moderate depression); 31-40 (severe depression); and >40 (extreme depression). Participants with symptom score of 0 were not included in the summary.
Time Frame: Month 3
Population: EITT population included any participant who received at least 1 dose of PTC589 and had a minimum of Month 3 assessment. 'Number analyzed' = participants with symptom score >1 for normal, mild, borderline, moderate, severe, or extreme depression. Data for a specific severity level was not collected if no evaluable participants were available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTC589
Number analyzed (Participants) | 40
units on a scale
  Normal: number analyzed (Participants) | 24
  Normal | 3.6 (2.41)
  Mild mood disturbance: number analyzed (Participants) | 9
  Mild mood disturbance | 13.1 (1.83)
  Borderline clinical depression: number analyzed (Participants) | 0
  Moderate depression: number analyzed (Participants) | 0
  Severe depression: number analyzed (Participants) | 0
  Extreme depression: number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Montgomery and Asberg Depression Rating Scale (MADRS) Total Score at Month 3
Description: The MADRS is a clinician-rated tool for measuring changes in depressive symptom severity. Ten core symptoms and cognitive features (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) were rated on a severity scale of 0 (no symptoms)) to 6 (symptoms of maximum severity). The total score was the sum of the scores on the 10 items, ranging from 0 to 60 with a higher score indicating increasing depressive symptoms.
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTC589
Number analyzed (Participants) | 40
units on a scale
  Baseline | 2.4 (2.60)
  Change at Month 3 | 0.1 (3.00)

9. Secondary Outcome: Change From Baseline in Time to Complete Time Up and Go (TUG) Test in ON State at Month 3
Description: Timed motor tests are simple, objective, quantitative measures for the assessment of Parkinson's disease. They include, in on-medication and off-medication state, timed recorded physical movements. Time Up and Go Test (TUG) is one of timed motor tests which is used to assess a person's mobility and requires both static and dynamic balance. This is a walking assessment. Participants start in the seated position, stand up, walk 7 meters, turn around, and sit back down. The entire process from leaving the chair to returning to the chair was timed. The total time was summarized under ON state with participants on dopamine therapy.
Time Frame: Baseline, Month 3
Population: EITT population included any participant who received at least 1 dose of PTC589 and had a minimum of the Month 3 assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PTC589
Number analyzed (Participants) | 18
seconds
  Baseline | 8.637 (1.8763)
  Change at Month 3 | -0.347 (1.1056)

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PTC589
Time Frame: 0 hour (predose) and 0.5, 1, 2, 4, 6, 8, and 12 hours postdose at Month 1 and 3
Population: as for outcome 9
Measure: Mean (Standard Error); unit: nanograms (ng)/milliliter (mL)
Arm/Group | PTC589
Number analyzed (Participants) | 23
nanograms (ng)/milliliter (mL)
  Month 1 | 3718.3 (311.6)
  Month 3 | 2903.5 (249.0)

11. Secondary Outcome: Level of Disease-Related Biomarker (Glutathione) in Plasma
Description: Glutathione lowest limit of quantification (LLOQ) = 0.01 micromoles (uM) and upper limit of quantification (ULOQ) = 27.83 uM in plasma.
Time Frame: Month 3
Population: EITT population included any participant who received at least 1 dose of EPI-589.
Measure: Mean (Full Range); unit: µM
Arm/Group | PTC589
Number analyzed (Participants) | 40
µM | 1.54 [0.37 to 8.33]

12. Secondary Outcome: Level of Disease-Related Biomarker (Glutathione) in Cerebrospinal Fluid (CSF)
Description: Glutathione LLOQ = 0.002 uM and ULOQ = 0.35 uM in CSF.
Time Frame: Month 3
Population: EITT population included any participant who received at least 1 dose of EPI-589. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Full Range); unit: µM
Arm/Group | PTC589
Number analyzed (Participants) | 36
µM | 0.10 [0.04 to 0.23]

13. Secondary Outcome: Level of Disease-Related Biomarker (Glutathione) in Urine
Description: Glutathione LLOQ = 0.01 uM, and ULOQ = 1.39 uM in urine.
Time Frame: Month 3
Population: EITT population included any participant who received at least 1 dose of EPI-589.
Measure: Mean (Full Range); unit: µM
Arm/Group | PTC589
Number analyzed (Participants) | 40
µM | 0.0000061 [0.00000034 to 0.000033]

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug (up to 4 months)
Description: Safety population included any participant who received at least 1 dose of PTC589.
Arm/Group | PTC589
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 29/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTC589 (N=41)
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 3
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 8
Abnormal sensation in eye (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Ocular discomfort (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Eructation (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Salivary hypersecretion (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Malaise (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Muscle strain (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Low density lipoprotein increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 2
Bradykinesia (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Hypogeusia (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT02462603/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT02462603/SAP_001.pdf